CLINICAL TRIAL: NCT01311284
Title: Comparison of Airtraq Nasotracheal Mcgrath and Macintosh Laryngoscope in Nasotracheal Intubation: A Manikin Study
Brief Title: Comparison Airway Devices in Nasotracheal Intubation in Manikin
Acronym: MGR-AR2010A1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manuel Ángel Gómez-Ríos (Other)
Responsible Party: Sponsor-Investigator, Manuel Ángel Gómez-Ríos, MD, Complexo Hospitalario Universitario de A Coruña
Organization: Complexo Hospitalario Universitario de A Coruña (Other)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: MGR-AR-2010-A1
Record Dates: First submitted 2011-03-07; First posted 2011-03-09 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Nasotracheal Intubation
Keywords: Nasotracheal intubation; Macintosh laryngoscope; Airtraq; McGrath; Manikin; airway management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Macintosh (Active Comparator)
  Interventions: Device: Macintosh laryngoscope, Airtraq NT, Mcgrath laryngoscope; Device: Macintosh laryngoscope
- Mcgrath (Active Comparator)
  Interventions: Device: Macintosh laryngoscope, Airtraq NT, Mcgrath laryngoscope; Device: McGrath
- Airtraq Nasotracheal (Active Comparator)
  Interventions: Device: Macintosh laryngoscope, Airtraq NT, Mcgrath laryngoscope; Device: Airtraq Nasotracheal

INTERVENTIONS:
Device: Macintosh laryngoscope, Airtraq NT, Mcgrath laryngoscope — Each participant will use the Macintosh laryngoscope (blade No. 3), laryngoscope Airtraq NT and Mcgrath Laryngoscope under conditions of normal and difficult airway in different simulated scenarios.
  Other Names: Macintosh; Airtraq NT; Mcgrath
Device: Macintosh laryngoscope — intubate with the macintosh laryngoscope
  Arms: Macintosh
Device: McGrath — Intubate with McGrath device
  Arms: Mcgrath
Device: Airtraq Nasotracheal — intubate with Airtraq Nasotracheal
  Arms: Airtraq Nasotracheal

SUMMARY:
Nasotracheal intubation is usually required in oral surgery to allow an unrestricted surgical approach. The standard method is generally performed using the Macintosh laryngoscope supported by Magill forceps. However, it is recommended to perform awake tracheal intubation in situations where a difficult airway is predicted, a scenario where this technique may be poorly tolerated by the patient. Although fibreoptic intubation is considered the "gold standard", sometimes it is difficult to perform and,therefore, alternatives are necessary. The hypothesis is that optical laryngoscopes as the Airtraq nasotracheal and Mcgrath can improve the time and/or success of nasotracheal intubation in a manikin.

ELIGIBILITY:
Inclusion Criteria:

* Be Component of service of anesthesiology C.H.U. A Coruña
* Give voluntary consent to participate in the study

Exclusion Criteria:

* Not meet the above criteria

Ages: 23 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2011-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Time in seconds required for a successful intubation attempt with the Macintosh laryngoscope, Airtraq NT and Mcgrath. | Two months

SECONDARY OUTCOMES:
Time visualization of the glottis | Two months
Intubation time | Two months
The duration of the first intubation attempt (whether successful or not) | Two months
Number of intubation attempts. | Two months
The success rate of placement of the endotracheal tube (ETT) in the trachea | Two months
Cormack and Lehane Grade | Two months
Number of operators needed | Two months
Severity of dental trauma | Two months
Satisfaction of the operators | Two months

CONTACTS AND LOCATIONS:
Locations (1):
- Complexo Hospitalario Universitario de A Coruña, A Coruña, A Coruña, Spain

REFERENCES:
- [Background] Hall CE, Shutt LE. Nasotracheal intubation for head and neck surgery. Anaesthesia. 2003 Mar;58(3):249-56. doi: 10.1046/j.1365-2044.2003.03034.x. PMID 12603455
- [Background] Gomez-Rios MA, Serradilla LN. Use of the Airtraq(R) optical laryngoscope for nasotracheal intubation in predicted difficult airway management in oral surgery. Can J Anaesth. 2010 Dec;57(12):1136-7. doi: 10.1007/s12630-010-9390-5. Epub 2010 Oct 2. No abstract available. PMID 20890692
- [Background] Lewis AR, Hodzovic I, Whelan J, Wilkes AR, Bowler I, Whitfield R. A paramedic study comparing the use of the Airtraq, Airway Scope and Macintosh laryngoscopes in simulated prehospital airway scenarios. Anaesthesia. 2010 Dec;65(12):1187-93. doi: 10.1111/j.1365-2044.2010.06514.x. Epub 2010 Oct 19. PMID 20958276
- [Background] Ueshima H, Asai T. Tracheal intubation in daylight and in the dark: a randomised comparison of the Airway Scope, Airtraq, and Macintosh laryngoscope in a manikin. Anaesthesia. 2010 Jul;65(7):684-7. doi: 10.1111/j.1365-2044.2010.06366.x. Epub 2010 May 28. PMID 20528836
- [Background] Lopez-Negrete IL, Salinas Aguirre U, Castrillo Villan JL, Rodriguez Delgado T, Colomino Alumbreros J, Aguilera Celorrio L. [Comparison of the view of the glottic opening through Macintosh and AirTraq laryngoscopes in patients undergoing scheduled surgery]. Rev Esp Anestesiol Reanim. 2010 Mar;57(3):147-52. doi: 10.1016/s0034-9356(10)70189-4. Spanish. PMID 20422847
- [Background] Liu L, Tanigawa K, Kusunoki S, Tamura T, Ota K, Yamaga S, Kida Y, Otani T, Sadamori T, Takeda T, Iwasaki Y, Hirohashi N. Tracheal intubation of a difficult airway using Airway Scope, Airtraq, and Macintosh laryngoscope: a comparative manikin study of inexperienced personnel. Anesth Analg. 2010 Apr 1;110(4):1049-55. doi: 10.1213/ANE.0b013e3181d2aad7. PMID 20357149
- [Background] McElwain J, Malik MA, Harte BH, Flynn NM, Laffey JG. Comparison of the C-MAC videolaryngoscope with the Macintosh, Glidescope, and Airtraq laryngoscopes in easy and difficult laryngoscopy scenarios in manikins. Anaesthesia. 2010 May;65(5):483-9. doi: 10.1111/j.1365-2044.2010.06307.x. Epub 2010 Mar 19. PMID 20337620
- [Background] Savoldelli GL, Schiffer E, Abegg C, Baeriswyl V, Clergue F, Waeber JL. Learning curves of the Glidescope, the McGrath and the Airtraq laryngoscopes: a manikin study. Eur J Anaesthesiol. 2009 Jul;26(7):554-8. doi: 10.1097/eja.0b013e3283269ff4. PMID 19522050
- [Background] Turkstra TP, Pelz DM, Jones PM. Cervical spine motion: a fluoroscopic comparison of the AirTraq Laryngoscope versus the Macintosh laryngoscope. Anesthesiology. 2009 Jul;111(1):97-101. doi: 10.1097/ALN.0b013e3181a8649f. PMID 19512871
- [Background] Savoldelli GL, Schiffer E, Abegg C, Baeriswyl V, Clergue F, Waeber JL. Comparison of the Glidescope, the McGrath, the Airtraq and the Macintosh laryngoscopes in simulated difficult airways*. Anaesthesia. 2008 Dec;63(12):1358-64. doi: 10.1111/j.1365-2044.2008.05653.x. PMID 19032306
- [Background] Ndoko SK, Amathieu R, Tual L, Polliand C, Kamoun W, El Housseini L, Champault G, Dhonneur G. Tracheal intubation of morbidly obese patients: a randomized trial comparing performance of Macintosh and Airtraq laryngoscopes. Br J Anaesth. 2008 Feb;100(2):263-8. doi: 10.1093/bja/aem346. PMID 18211999
- [Background] Maharaj CH, Costello JF, Harte BH, Laffey JG. Evaluation of the Airtraq and Macintosh laryngoscopes in patients at increased risk for difficult tracheal intubation. Anaesthesia. 2008 Feb;63(2):182-8. doi: 10.1111/j.1365-2044.2007.05316.x. PMID 18211450
- [Background] Maharaj CH, Buckley E, Harte BH, Laffey JG. Endotracheal intubation in patients with cervical spine immobilization: a comparison of macintosh and airtraq laryngoscopes. Anesthesiology. 2007 Jul;107(1):53-9. doi: 10.1097/01.anes.0000267529.71756.f0. PMID 17585215
- [Background] Maharaj CH, O'Croinin D, Curley G, Harte BH, Laffey JG. A comparison of tracheal intubation using the Airtraq or the Macintosh laryngoscope in routine airway management: A randomised, controlled clinical trial. Anaesthesia. 2006 Nov;61(11):1093-9. doi: 10.1111/j.1365-2044.2006.04819.x. PMID 17042849
- [Background] Maharaj CH, Costello JF, Higgins BD, Harte BH, Laffey JG. Learning and performance of tracheal intubation by novice personnel: a comparison of the Airtraq and Macintosh laryngoscope. Anaesthesia. 2006 Jul;61(7):671-7. doi: 10.1111/j.1365-2044.2006.04653.x. PMID 16792613
- [Background] Maharaj CH, Higgins BD, Harte BH, Laffey JG. Evaluation of intubation using the Airtraq or Macintosh laryngoscope by anaesthetists in easy and simulated difficult laryngoscopy--a manikin study. Anaesthesia. 2006 May;61(5):469-77. doi: 10.1111/j.1365-2044.2006.04547.x. PMID 16674623
- [Background] Maharaj CH, Costello J, Higgins BD, Harte BH, Laffey JG. Retention of tracheal intubation skills by novice personnel: a comparison of the Airtraq and Macintosh laryngoscopes. Anaesthesia. 2007 Mar;62(3):272-8. doi: 10.1111/j.1365-2044.2007.04938.x. PMID 17300305
- [Background] Maassen R, Lee R, Hermans B, Marcus M, van Zundert A. A comparison of three videolaryngoscopes: the Macintosh laryngoscope blade reduces, but does not replace, routine stylet use for intubation in morbidly obese patients. Anesth Analg. 2009 Nov;109(5):1560-5. doi: 10.1213/ANE.0b013e3181b7303a. Epub 2009 Aug 27. PMID 19713258
- [Background] Ray DC, Billington C, Kearns PK, Kirkbride R, Mackintosh K, Reeve CS, Robinson N, Stewart CJ, Trudeau T. A comparison of McGrath and Macintosh laryngoscopes in novice users: a manikin study. Anaesthesia. 2009 Nov;64(11):1207-10. doi: 10.1111/j.1365-2044.2009.06061.x. PMID 19825056
- [Background] Walker L, Brampton W, Halai M, Hoy C, Lee E, Scott I, McLernon DJ. Randomized controlled trial of intubation with the McGrath Series 5 videolaryngoscope by inexperienced anaesthetists. Br J Anaesth. 2009 Sep;103(3):440-5. doi: 10.1093/bja/aep191. Epub 2009 Jul 15. PMID 19605408